CLINICAL TRIAL: NCT05203458
Title: HER2 Retrospective Epidemiology Study Prevalence and Clinicopathologic Features of Different HER2 Level in Chinese Breast Cancer Patients (HER2 PATH)
Brief Title: Prevalence and Clinicopathologic Features of Different HER2 Level in Chinese Breast Cancer Patients
Acronym: HER2 PATH
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9673R00011
Record Dates: First submitted 2021-10-20; First posted 2022-01-24 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer, HER2
Keywords: breast cancer,HER2
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective study aims to estimate the prevalence of different HER2 expression levels (HER2+, HER2-low, HER2 Ø) in approximately 200 breast cancer patients at FUSCC through the year of 2015 and 3000 breast cancer patients from about 10 medical centres in China between July 2021 and July 2022

DETAILED DESCRIPTION:
This is a multicenter, retrospective study to estimate the prevalence of different HER2 expression levels (HER2+, HER2-low, HER2 Ø) in approximately 200 breast cancer patients at FUSCC through the year of 2015 and 3000 breast cancer patients from about 10 medical centres in China between July 2021 and July 2022.

This study will be divided into two parts： The first part will include 200 subjects who were pathologically diagnosed with breast cancer at FUSCC between Jan 2015 and Dec 2015 (PART 1).This part will collect rescored HER2 expression level results based on the archived HER2 IHC slides and re-staining and re-scoring HER-2 IHC while relative demographic, treatment, and clinicopathologic data will be extracted from the FUSCC Breast Cancer Single Disease Database.

The second part will include 3000 patients from all sites in China who were pathologically diagnosed with breast cancer between July 2021 and July 2022 (PART 2). This part will collect re-assessed HER2 expression level results based on the archived HER2 IHC slides. The general information of patients, diagnosis, clinicopathological information were collected from medical records, Hospital Information System (HIS) and Laboratory Information Management System (LIS).

In PART 2, among 3000 patients, 270 from all participating sites except FUSCC should have enough tumor tissue for re-staining and re-scoring HER-2 IHC at FUSCC to analyse the concordance between leading site and other centers.

In PART 2, among 3000 patients, 800 HER-2 IHC samples will be selected for the validation through AI-assisted HER2 assessment system

ELIGIBILITY:
Inclusion Criteria:

Patients fulfilling all of the following criteria will be eligible for this study:

* Male and female patients must have a histological confirmed diagnosis of BC
* The patients must be ≥18 years old at the diagnosis.
* In PART 1, all patients should be diagnosed at FUSCC between Jan 2015 and Dec 2015.
* In PART 2, all patients should be diagnosed at all participating sites between July 2021 and July 2022.
* Provision of at least 1 archived HER2 IHC slides associated with confirmed diagnosis of BC, which are in good condition for rescoring.
* FISH result is available for HER2 IHC2+ in primary scoring.

Exclusion Criteria:

Patients who meet any of the following criteria will be disqualified from entering the study:

* Absence of all demographic, histopathologic, clinicopathologic information .
* Have a history of other malignancies, other than basal cell carcinoma of the skin and squamous cell carcinoma of the skin.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 3000 eligible breast cancer patients from about 10 medical sites in China from July 2021 to July 2022 and 200 patients admitted at FUSCC from January 1st 2015 to December 31st 2015. Eligible patients will be those who had qualified archived HER2 IHC slides.
Sampling Method: Probability Sample
Enrollment: 3136 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
The Prevalence of different HER2 expression levels | Within one year
  To estimate the prevalence of different HER2 expression levels (HER2+, HER2-low(defined as IHC 1+,2+/ISH-), HER2 Ø) in Chinese breast cancer patients in PART 2.

SECONDARY OUTCOMES:
Tumor size of histopathological | Within one year
  Tumor size of Histopathological characteristic by different HER2 expression level (Ø /Low/High) in PART 1 and PART 2
Positive lymph node number of the histopathological | Within one year
  Positive lymph node number of histopathological characteristic by different HER2 expression level (Ø /Low/High) in PART 1 and PART 2
TNM stage by different HER2 expression levels | Within one year
  TNM stage by different HER2 expression level (Ø /Low/High) in PART 1 and PART 2
Pathological type of histopathological | Within one year
  Pathological type by different HER2 expression level (Ø /Low/High) in PART 1 and PART 2
Histological grade of histopathological | Within one year
  Histological grade by different HER2 expression level (Ø /Low/High) in PART 1 and PART 2
Multi-focal of histopathological | Within one year
  Multi-focal by different HER2 expression level (Ø /Low/High) in PART 1 and PART 2
ER status of histopathological | Within one year
  ER status by different HER2 expression level (Ø /Low/High) in PART 1 and PART 2
ER percentage by different HER2 expression levels. | Within one year
  ER percentage by different HER2 expression level (Ø /Low/High) in PART 1 and PART 2
PR status of histopathological | Within one year
  PR status by different HER2 expression level (Ø /Low/High) in PART 1 and PART 2
PR percentage by different HER2 expression levels. | Within one year
  PR(Progesterone Receptor) percentage by different HER2 expression level (Ø /Low/High) in PART 1 and PART 2
Ki-67 percentage by different HER2 expression levels. | Within one year
  Histopathological and clinicopathological characteristics by different HER2 expression level (Ø /Low/High) including: Ki-67 percentage,in PART 1 and PART 2
HER2 IHC score of histopathological | Within one year
  HER2 IHC score by different HER2 expression level (Ø /Low/High) in PART 1 and PART 2
FISH status of histopathological | Within one year
  FISH status by different HER2 expression level (Ø /Low/High) in PART 1 and PART 2
The concordance between historical scoring and reassess scoring in each IHC score category (IHC score Ø, 1+, 2+and 3+) | Within one year
  To estimate the concordance between historical scoring and reassess scoring in each IHC score category (IHC score Ø, 1+, 2+and 3+) in PART 2
The concordance of HER2 expression between manual and AI assisted HER2 interpretation | Within one year
  To estimate the concordance of HER2 expression between manual and AI assisted HER2 interpretation among 800 patients in PART 2
The concordance of HER2 expression between leading site (FUSCC) and other centers | Within one year
  To estimate the concordance of HER2 expression between leading site (FUSCC) and other centers among 270 patients in PART 2

OTHER OUTCOMES:
The prevalence of HER2 IHC0 and HER2 IHC >0<1+ | Within one year
  To estimate the prevalence of HER2 IHC0 and HER2 IHC >0<1+ in PART 2
Age at diagnosis of patients' demographic at baseline | At baseline
  Age at diagnosis of patients' demographic at baseline by different HER2 expression level in PART 1
BMI of patients' demographic at baseline | At baseline
  BMI of patients' demographic at baseline by different HER2 expression level in PART 1
Menopause or not of patients' demographic at baseline | At baseline
  Menopause or not of patients' demographic at baseline by different HER2 expression level in PART 1
The baseline treatment patterns across patients with different HER2 expression levels | At baseline
  Patients' treatment patterns at baseline, by different HER2 expression level in PART 1

CONTACTS AND LOCATIONS:
Overall Officials: Wentao Yang, Dr., Principal Investigator — Fudan University
Locations (7):
- China (7):
  - Research Site, Shanghai, Shanhai
  - Research Site, Guangzhou
  - Research Site, Jinan
  - Research Site, Shenyang
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lv H, Yue J, Zhang Q, Xu F, Gao P, Yang H, Nie X, Kong L, Zhang G, Li J, Xiao S, Wu H, Xing A, Hong M, Fan J, Guan H, Cao P, Ni H, Yang W. Prevalence and concordance of HER2-low and HER2-ultralow status between historical and rescored results in a multicentre study of breast cancer patients in China. Breast Cancer Res. 2025 Mar 25;27(1):45. doi: 10.1186/s13058-025-02001-0. PMID 40134013
- See also: redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9673R00011&attachmentIdentifier=3957d0f6-36a1-45a9-91ec-13eda815e3d2&fileName=D9673R00011_HER2_PATH_CSR__synopsis.pdf&versionIdentifier=